CLINICAL TRIAL: NCT04308200
Title: The Effect of the Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach for Children With Cerebral Palsy: a Randomized Controlled Trial
Brief Title: The Effect of the CO-OP Approach for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZEYNEP KOLİT (Other)
Responsible Party: Sponsor-Investigator, ZEYNEP KOLİT, Principal Investigator, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 18/624
Record Dates: First submitted 2020-03-05; First posted 2020-03-13 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Cerebral Palsy; Cognitive Orientation
Keywords: Cerebral Palsy; Cognitive Orientation; occupations; functional status
MeSH Terms: conditions — Cerebral Palsy; Orientation, Spatial

STUDY DESIGN:
Intervention Model Description: The study was a single blinded and randomized controlled trial. All children included in the study were evaluated by a single evaluator who was blind to therapy at baseline and at the end of treatment. The study was completed with a total of 30 individuals, 15 in the CO-OP+ neurodevelopmental therapy (NDT) and 15 in the NDT group. Both groups received NDT for 45 minutes once daily, two times a week for period of 6 weeks by the same physiotherapist. The NDT protocol is improving muscular tone and movement patterns. All sessions incorporated handling techniques that aimed to alter muscle tone during movement and to facilitate anti-gravity and postural reactions. All children who met the inclusion criteria using GMFCS and MACS were evaluated with sociodemographic data, activity daily log, COPM and PEDI. The CO-OP group received twelve sessions of intervention, with the baseline and end of treatment assessments, each lasting approximately one hour.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO-OP+NDT group (Other): The CO-OP+NDT group received twelve sessions of CO-OP approach, with the baseline and end of treatment assessments, each lasting approximately one hour. Parents and / or caregivers were advised to observe sessions as often as possible to encourage adaptation and transfer to life. Furthermore, CO-OP+NDT group received NDT for 45 minutes once daily, two times a week for period of 6 weeks by the same physiotherapist.
  Interventions: Other: CO-OP approach; Other: NDT
- NDT group (Other): NDT group received just NDT for 45 minutes once daily, two times a week for period of 6 weeks by the same physiotherapist. The NDT protocol is improving muscular tone and movement patterns. All sessions incorporated handling techniques that aimed to alter muscle tone during movement and to facilitate anti-gravity and postural reactions.
  Interventions: Other: NDT

INTERVENTIONS:
Other: CO-OP approach — There are 3 stages in the CO-OP approach. Stage I, the Preparation Stage, is primarily concerned with establishing the "goal". Before the first interview, the child was contacted, the family and the child were informed, and it was checked whether they met the prerequisites. At this stage, 3 targets were selected and the basic performance level was determined. Stage II, the Acquisition Stage, is essentially the "plan" and "do" stage, in which the work of using strategies to acquire skills is done. This stage originally comprised 10 sessions. At this stage, the first session enabling principles were implemented and the global strategy "goal-plan-do-check" was introduced. The family attended this process with observation. Parents / caregivers were encouraged to make observations to generalize strategies. Stage III, the Verificatíon stage usually consists of only one session in which "control" is performed; the progress made was revised as learned strategies.
  Arms: CO-OP+NDT group
Other: NDT — All participations received NDT for 45 minutes once daily, two times a week for period of 6 weeks by the same physiotherapist. The NDT protocol is improving muscular tone and movement patterns. Although the treatment activities varied for each CP participant, the overall goals (improved smoothness and efficiency of movement), which included improved trunk, hip, knee and ankle control, were the same for all CP participants. All sessions incorporated handling techniques that aimed to alter muscle tone during movement and to facilitate anti-gravity, weight-shifting and postural reactions.

SUMMARY:
In the literature, despite the reported positive findings of the Cognitive Orientation to daily Occupational Performance (CO-OP) approach, studies in this area have been limited and it is stated that studies involving more sample groups are needed (24-27). In addition, no studies investigating the effect of the CO-OP approach on functional status were found. The purpose of this study was to investigate the effects of CO-OP approach in terms of occupational performance and satisfaction also functional status in children with cerebral palsy (CP) and to determine parents' satisfaction level from CO-OP.

The hypotheses of the study are: The CO-OP approach has no effect on occupational performance in children with CP. CO-OP approach has no effect on occupational satisfaction in children with CP. The CO-OP approach has no effect on the functional status of children with CP.

DETAILED DESCRIPTION:
Statistical analyses were performed using the Statistical Package for the Social Sciences (SPSS) version 22 (IBM SPSS Statistics; IBM Corporation, Armonk, NY). One sample Kolmogorov-Smirnov Test was used evaluate the distribution of variables prior to test selection. Group characteristics and outcome measures are described using mean and standard deviations for continuous variables and frequencies and proportions for categorical variables. Descriptive statistics were presented as median for the non-normally distributed quantitative and ordinal data and number (percentage) for the categorical variables. Differences in continuous variables (age, education, BMI, duration of diagnosis,) among groups were analyzed with the Mann Whitney U. Statistical differences in COPM and PEDI scores between baseline and post-treatment was analyzed with "Wilcoxon's signed-rank test" within groups. The z-score obtained from the Wilcoxon signed-rank test was reported to present a standardized measure of the difference between the mean ranks of the negative and positive groups. Comparison of changes between groups were analyzed with "Mann-Whitney U" test for COPM and PEDI scores. Statistical significance level was assumed at p<0.05.

Clinical significance was calculated by using the Cohen d effect size index in independent groups. Clinical significance was determined according to Cohen's recommended limit values (0,2 small; 0,5 moderate and 0,8 large effect).

ELIGIBILITY:
Inclusion Criteria:

* being between 5-12 years of age
* being diagnosed with CP
* being at level I, II, or III according to the Gross Motor Function Classification Scale (GMFCS)
* being at level I, or II according to the Manual Ability Classification System (MACS)
* having experienced motor performance problems in daily activities, as reported by parents and/or children during interview; have sufficient language ability to communicate with and be understood during treatment.

Exclusion Criteria:

* receiving another treatment other than NDT
* being diagnosed with mental retardation
* having serious visual or hearing problems.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | It was re-applied 5 weeks after the baseline evaluations were made.
  The COPM was used in this study to establish goals for each child prior to intervention. It is a semi-structured interview designed to help clients identify occupational performance issues and priorities in the areas of self-care, productivity (school), and leisure, in which they have difficulty performing. In this study, children and their parents selected the "training goals" collaboratively by rating on a 10-point scale displaying their goals in terms of satisfaction and performance. The children and their parents scored the COPM independently before and after intervention based on goals set by the child and supported by the parents. Changes in performance and satisfaction scores before and after intervention were determined separately. A change score of two points or more on the COPM is considered clinically significant
Pediatric Evaluation of Disability Inventory (PEDI) | It was re-applied 5 weeks after the baseline evaluations were made.
  PEDI is a clinical measurement tool developed by Haley et al to evaluate the functional status of children. In particular, it is arranged to determine the functions of young children . It can also be used for older children whose functional performance falls below that expected for 7.5- year-old normally developing children. PEDI consists of three main sections, functional skills, caregiver assistance and modifications. Each of these sections evaluates the areas of self-care, mobility and social function. Each of the PEDI subsections can be used separately.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | It was applied to the caregivers of the CO-OP + NDT group within 1 days after 5 weeks of training.
  It is a reliable, easily applicable assessment tool that is accepted in the world literature. VAS is used to convert some non-quantifiable values into numeric data. It is the scale in which a person marks his / her current emotion level with a vertical line on a 10 cm scale. Every emotion is evaluated between the fact that the feeling is never experienced and that it is being experienced completely. Post-intervention satisfaction levels of the parents in the CO-OP group were determined using VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Kolit, MSc, Principal Investigator — Hacettepe University; Gamze Ekici Çağlar, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No